CLINICAL TRIAL: NCT02371512
Title: A Multicenter, Randomized, Controlled Study to Assess Mitral vAlve reconsTrucTion for advancEd Insufficiency of Functional or iscHemic ORigiN
Acronym: MATTERHORN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: The Clinical Trials Centre Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MATTERHORN
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Mitral Valve Insufficiency
Keywords: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous mitral valve repair (MitraClip system ) (Experimental): Percutaneous mitral valve repair (simultaneous left atrial and ventricular pressure assessment suggested) with MitraClip system (Abbott)
  Interventions: Device: MitraClip system (Abbott Vascular, Menlo Park, USA)
- Mitral valve surgery (Active Comparator): Mitral valve surgery or mitral valve replacement (technique and access at the discretion of the participating surgical center, MACE procedure and tricuspid annuloplasty possible)
  Interventions: Procedure: Mitral valve surgery

INTERVENTIONS:
Device: MitraClip system (Abbott Vascular, Menlo Park, USA) — Valve repair with the MitraClip system (Abbott Vascular, Menlo Park, USA) consists of a steerable guide through which a Clip Delivery System is advanced to the left atrium.
  Arms: Percutaneous mitral valve repair (MitraClip system )
Procedure: Mitral valve surgery — Mitral valve surgery or mitral valve replacement (technique and access at the discretion of the participating surgical center, MACE procedure and tricuspid annuloplasty possible)
  Arms: Mitral valve surgery

SUMMARY:
Study to assess mitral valve therapy for advanced insufficiency of functional or ischemic origin in patients with moderate-to-severe mitral regurgitation (MR) of primarily functional pathology and reduced left ventricular function considered to be at high surgical risk

DETAILED DESCRIPTION:
Secondary or functional mitral regurgitation (MR) results from a geometrical distortion of a dysfunctional left ventricle leading to tethering of mitral valve leaflets by papillary muscle displacement, annular dilatation and/or reduced closing forces in a structurally normal mitral valve. It occurs in over 30% of patients with systolic heart failure. Despite optimal medical care it is associated with increased mortality and hospitalization rates leaving elimination of MR as the only therapeutic option. Nevertheless, traditionally, mitral valve surgery has been the therapy of choice in this setting.

As mitral valve surgery has so far been only investigated in retrospective single center registries, which have shown conflicting results. it has a class IIb recommendation, level of evidence C, in these patients without indication for coronary revascularization in the current guidelines of the European Society of Cardiology. In recent years percutaneous mitral valve repair with the MitraClip (PMVR) has evolved as an important therapeutic option in this type of patient with widespread use particularly in Europe, where the device was CE-marked in 2008. PMVR has been compared to mitral valve surgery (repair and replacement) in the randomized, controlled EVEREST II trial in patients with primary MR, which were good candidates for surgery, and was shown to be less effective than surgery in this context. However, no randomized, controlled data are available comparing PMVR and mitral valve surgery in patients with depressed left ventricular function and secondary MR, who have a considerably higher perioperative risk than the EVEREST II population. Like mitral valve surgery it has a class IIb, level of evidence C, recommendation in current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant mitral regurgitation of primarily functional pathology
* Left Ventricular Ejection Fraction (LVEF) ≥20% determined by echocardiography
* High surgical risk as determined by Heart Team consensus
* Documented New York Heart Association Class II to Class IV heart failure, despite optimal standard of care therapy
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Echocardiographic evaluation not available or not suitable for analysis at baseline
* Severe tricuspid regurgitation according to current guidelines5
* Other severe valve disorders requiring intervention according to current
* Coronary revascularization or cardiac resynchronization (CRT) device implantation within 1 month before the procedure
* Patient not amenable for mitral valve surgery/ percutaneous mitral valve reconstruction as judged by Heart Team
* Key information from patients (e.g. NYHA, MR grade) not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Composite of death, rehospitalisation for heart failure, reintervention (repeat operation or repeat intervention), assist device implantation and stroke (whatever is first) 12 months post intervention; equivalently "freedom from event" | 12 months post intervention
  Composite of death, rehospitalisation for heart failure, reintervention (repeat operation or repeat intervention), assist device implantation and stroke (whatever is first) 12 months post intervention; equivalently "freedom from event"

SECONDARY OUTCOMES:
Recurrence of grade 3 or 4 mitral regurgitation within 12 months post intervention | 12 months post intervention
  Recurrence of grade 3 or 4 mitral regurgitation within 12 months post intervention
Change in 6 Minute Walk Test distance from baseline to 12 month post intervention (difference "12 months minus baseline | 12 months post intervention
  Change in 6 Minute Walk Test distance from baseline to 12 month post intervention (difference "12 months minus baseline
Change in NYHA functional class from baseline to 12 months post intervention | 12 months post intervention
  Change in NYHA functional class from baseline to 12 months post intervention
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) score from baseline to 12 months post intervention | 12 months post intervention
  Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) score from baseline to 12 months post intervention
Echocardiographic assessment of left ventricular remodelling | 12 months post intervention
Change in serum BNP from baseline to 12 months post intervention | 12 months post intervention
Length of stay ICU / hospital | Participants will be followed for the duration of hospital stay, an expected average of 1 week. However, in some patients the hospital stay can be exceed this time frame, when complications occur.
Number of patients in whom operative or interventional mitral valve repair can not be performed (need for mitral valve replacement) | 12 months post intervention
  The primary therapeutic strategy should be a repair of the study. For patients undergoing interventional therapy this endpoint is reached if the clip procedure is aborted and a mitral valve replacement is performed. In patients undergoing surgery the endpoint is reached if the surgeon decides to implant a mitral valve during the same procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Baldus, Prof. Dr. med., Study Director — Herzzentrum Uniklinik Köln
Locations (1):
- Heart Center University of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Baldus S, Doenst T, Pfister R, Gummert J, Kessler M, Boekstegers P, Lubos E, Schroder J, Thiele H, Walther T, Kelm M, Hausleiter J, Eitel I, Fischer-Rasokat U, Bufe A, Schmeisser A, Ince H, Lurz P, von Bardeleben RS, Hagl C, Noack T, Reith S, Beucher H, Reichenspurner H, Rottbauer W, Schulze PC, Muller W, Frank J, Hellmich M, Wahlers T, Rudolph V; MATTERHORN Investigators. Transcatheter Repair versus Mitral-Valve Surgery for Secondary Mitral Regurgitation. N Engl J Med. 2024 Nov 14;391(19):1787-1798. doi: 10.1056/NEJMoa2408739. Epub 2024 Aug 31. PMID 39216093